CLINICAL TRIAL: NCT05060939
Title: Characterization of the Viral Genome and Humoral Immune Response in COVID-19 Vaccinated Patients With SARS-CoV-2 Infection
Brief Title: SARS-CoV-2 Infection in COVID-19 Vaccinated Patients
Acronym: COVID-IVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL21_0748
Record Dates: First submitted 2021-09-28; First posted 2021-09-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: SARS-CoV-2, COVID-19; vaccine,; variant; host-immune response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: COVID-19 vaccinated people — Patients with at least one dose of COVID-19 vaccine tested for SARS-CoV-2 infection with RT-PCR on respiratory specimen. RT-PCR, serological testing and viral sequencing will be applied on patient's samples

SUMMARY:
Vaccination of the population is crucial in the fight against the COVID-19 pandemic. Although most available vaccines have an estimated efficacy against symptomatic infection of 65-95%, this can be significantly reduced if the patient has co-morbidities such as immunosuppression or if the full vaccination schedule is not followed. Infection with SARS-CoV-2 variants, carrying mutations, notably on the spike protein, may also be associated with escape from immunity acquired by vaccination. Indeed, in vitro studies have shown a decrease in sensitivity to neutralizing antibodies acquired after vaccination or even after infection for certain variants such as variant B.1.351 (beta variant according to the WHO, first detection in South Africa) or variant B.1.617.2. (delta variant according to the WHO, first detection in India). On the other hand, cases of COVID-19 following a full vaccination regimen have recently been reported. With the increasing detection of new variants and in the context of increasing vaccination coverage of the population, one of the priority missions of the National Reference Centre (NRC) for respiratory infection viruses is to clinically and virologically investigate all cases of infection in vaccinated patients. The main objective is to determine whether a particular variant is over-represented in vaccinated patients with an infection. The secondary objective is to study the humoral immune response in COVID-19 vaccinated patients with and without SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* Persons having given their written consent and accepting a follow-up every 6 months for 24 months, followed by a final visit at 36 months.
* Persons affiliated to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

- Pregnant or lactating woman

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Distribution of the clade and lineage of SARS-CoV-2 in vaccinated patients | At inclusion
  Whole genome sequencing of SARS-CoV-2 RT-PCR positive samples

SECONDARY OUTCOMES:
Titers of SARS-CoV-2 antibodies | At inclusion
  Measurement of anti-N, anti-S antibody titers with commercial serological tests.
  Measurement of neutralizing antibody titers with virus neutralization assay
Titers of SARS-CoV-2 antibodies | At inclusion
  Neutralizing antibody titer measurements for different variants including graded variants of concern by Public Health France.
Titers of SARS-CoV-2 antibodies | At inclusion
  Measurement of interferon gamma titer by an ELISA method after stimulation with a peptide immunogenic

CONTACTS AND LOCATIONS:
Locations (1):
- BAL Antonin, Lyon, National Reference Center For Respiratory Viruses, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy A, Saade C, Josset L, Clement B, Morfin F, Destras G, Valette M, Icard V, Billaud G, Oblette A, Debombourg M, Garrigou C, Brengel-Pesce K, Generenaz L, Saker K, Hernu R, Pozzetto B, Lina B, Trabaud MA, Trouillet-Assant S, Bal A. Determinants of protection against SARS-CoV-2 Omicron BA.1 and Delta infections in fully vaccinated outpatients. J Med Virol. 2023 Aug;95(8):e28984. doi: 10.1002/jmv.28984. PMID 37503561